CLINICAL TRIAL: NCT05785936
Title: Impact of Desensitization Therapies on the Immune Response of Highly Sensitized Patients Awaiting Kidney Transplantation
Brief Title: Immune Response in Desensitized Patients
Acronym: DELIGHT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Principal Investigator, Noble_Johan, MD, Principal investigator, University Hospital, Grenoble
Other Study IDs: 2022-A02445-38
Record Dates: First submitted 2023-03-09; First posted 2023-03-27 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Kidney Transplant Rejection
Keywords: HLA sensitization; Desensitization; Antibody secreting cells
MeSH Terms: interventions — Desensitization, Psychologic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood for PBMC (peripheral mononuclear cells) Medullary samples Lymph node samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Highly sensitized and desensitized kidney transplanted group: Patient that were HLA desensitized for kidney transplantation
  Interventions: Procedure: Desensitization
- Highly sensitized and non-desensitized kidney transplanted group: Patient that were not HLA desensitized for kidney transplantation but were highly sensitized and received a kidney graft due to local priority system
- Healthy donors

INTERVENTIONS:
Procedure: Desensitization — Patients that received apheresis and anti-cluster of differentiation antigen 20 for desensitization priori to kidney transplantation
  Groups: Highly sensitized and desensitized kidney transplanted group

SUMMARY:
Kidney transplantation is the best treatment for chronic renal failure in terms of morbidity and mortality, quality of life for patients and health economics. Sensitization with anti-Human Leukocyte Antigen antibodies is a barrier to access to transplantation.

Highly-sensitized patients wait 2 to 3 times longer on the waiting list with important health and economic consequences. Desensitization strategies by apheresis techniques allow access to a transplant with a negative crossmatch (absence of specific HLA antibodies against their donor) on the day of the transplant.

The main objective of this study is to assess the impact of desensitization on the antibody memory immune response in highly sensitized patients awaiting kidney transplantation.

The analyses will be based on samples from the 20 patients (10 desensitized transplanted patients, 5 highly sensitized non-desensitized transplanted patients and 5 healthy donors) at the University Hospital of Grenoble, France.

Analyses will include phenotypic and immuno-metabolic analysis by flow cytometry of antibody-secreting cells, a functional analysis by anti HLA ELISpot B technique and histological analysis of post-kidney transplantation follow-up renal biopsies with gene expression mapping (RNA tissue labeling using the Nanostring technique) within the renal parenchyma.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age >18 years) with end-stage renal disease (on hemodialysis or peritoneal dialysis or stage V chronic kidney disease) who are candidates for pre-renal transplantation desensitization from living or deceased donors.
* For women of childbearing age: a plasma pregnancy test before inclusion is mandatory. Highly effective contraception for women of childbearing age is required throughout the study period:
* combined hormonal contraception (containing estrogen and progestin)
* contraception associated with ovulation inhibition :

  * oral
  * intravaginal
  * transdermal
* Progestin-only hormonal contraception associated with ovulation inhibition:

  * oral
  * injectable
  * implantable
* intrauterine device (IUD) - intrauterine hormone delivery system (IUS)
* bilateral tubal occlusion
* vasectomized partner
* sexual abstinence
* Have signed the DELIGHT protocol consent.
* Affiliated to a social security system
* Can be contacted in case of emergency
* For the control groups :
* Healthy controls from blood samples (centrifugation ring) from the French Blood Agency. The use of healthy controls is necessary to compare immunological analyses to a reference group without immunosuppression.
* Highly sensitized kidney transplant patients without the need for de-immunization. Hyperimmunization is defined by a Panel Reactive Antibody score > 85%. Transplantation can be from deceased or living donors.

Exclusion Criteria:

* Patients who object to the use of their data and/or samples in the research
* Patients having received an immunosuppressive treatment in the 12 months preceding the inclusion
* All protected persons: pregnant women, parturients, nursing mothers, persons deprived of liberty by judicial or administrative decision, persons under legal protection.
* Subjects in a period of exclusion from another study
* Subject under administrative or judicial supervision
* Subject unable to be contacted in case of emergency

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 15 highly sensitized patients: 10 that received desensitization before kidney transplan tation and 5 that were not desensitized before kidney transplantation.
  5 healthy donors
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Flow Cytometry analyses of Peripheral Blood Mononuclear Cells | Before desensitization, at the time of transplantation and Before desensitization, at the time of transplantation and post transplantation
  Change of the percentage of "antibody secreting cells" (plasmablasts) over time
Change in Anti HLA B-cell ELISpot response | Before desensitization, at the time of transplantation and Month 3, Month 6 and Month 12 post transplantation
  Change in the number of Spot over time
Change in Flow Cytometry analyses of medullary cells | The first day of desensitization and at the day of kidney transplantation
  Change in the percentage of "antibody secreting cells" (plasmablasts) over time
Change in analyses of RNA expression on renal histology | Month1, Month 3 and Month 12 post transplantation
  CHange in percentage of gene expression using Nanostring technology